CLINICAL TRIAL: NCT06124443
Title: Maternal Diabetes as a Risk Factor for Congenital Heart Defects in Infants of Diabetic Mothers.
Brief Title: Congenital Heart Defects
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moustafa Adel Mohamed Ahmed, 71515,Assiut, Assiut University
Other Study IDs: Congenital heart defects
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Infants & children of diabetic mothers
- Controls: Infants & children of non-diabetic mothers

SUMMARY:
Describe the relationship between maternal diabetes and congenital heart defects in infants born to diabetic mothers referred to NICU unit & Outpatient clinics of Assiut University Childeren's hospital.We will compare between 2 groups. Cases will represent infants of diabetic mothers & Conteols will represent infants of non-diabetic mothers.

DETAILED DESCRIPTION:
Congenital heart disease is defined as a gross structural abnormality of the heart or intra-thoracic great vessels that is actually or potentially of functional significance .The prevalence of CHD at birth has been relatively variable at 4.05 to 10.4 cases per 1000 live births in different surveys however,it is 5.0% in infants of diabetic mothers (IDMs).CHD is the most common congenital problem in children accounting for nearly 25% of all congenital malformations .CHDs are one of the significant causes of infant morbidity and mortality. Gestational diabetes mellitus (GDM) is the most common medical complication of pregnancy. It is associated with maternal and neonatal adverse outcomes. Maintaining adequate blood glucose levels in GDM reduces morbidity for both mother and baby. Pregnancy is associated with insulin resistance (IR) and hyperinsulinemia that may predispose some women to develop diabetes. Gestational diabetes has been defined as any degree of glucose intolerance with an onset, or first recognition during pregnancy. Diabetes during pregnancy could be a de novo that arises during pregnancy for the first time and could disappear or persist after delivery (gestational DM) or could start as pre-gestational, before the onset of pregnancy. The incidence of impaired glucose tolerance in pregnancy ranges between 3-10% and varies according to the average incidence of diabetes in the general Population. Specific CHDs that are more commonly seen in IDMs include ventricular septal defect (VSD), transposition of the great arteries (TGAs), and aortic stenosis (AS).Approximately one third of neonates with CHD require intervention in the first month of life . Clinical manifestation of CHD varies according to the type of lesion. Neonates with respiratory distress , cyanosis, feeding difficulties, and low cardiac output are common presentations of CHD . So diagnosis of CHD at the earliest possible time is very important as early referral and appropriate intervention in some of these cases are lifesaving.

ELIGIBILITY:
Inclusion Criteria:

The study will include infants of diabetic mothers and infants of non-diabetic mothers not previously screened for congenital heart defects.

Exclusion Criteria:

Other risk factors for congenital heart defects including congenital infections like TORCH infection, teratogenic drugs ( lithium or isotretinoin), , alcohol, or smoking.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Neonates and children of diabetic and non-diabetic mothers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Assesment of prevalence of congenital heart defects among infants of diabetic mother compared to that in infants of non-diabetic mothers. | Baseline
  Assesment of prevalence of congenital heart defects among infants of diabetic mother compared to that in infants of non-diabetic mothers.

REFERENCES:
- [Background] Al-Biltagi M, Tolba OA, Rowisha MA, Mahfouz Ael-S, Elewa MA. Speckle tracking and myocardial tissue imaging in infant of diabetic mother with gestational and pregestational diabetes. Pediatr Cardiol. 2015 Feb;36(2):445-53. doi: 10.1007/s00246-014-1033-0. Epub 2014 Oct 7. PMID 25287219
- [Background] Classification and diagnosis of diabetes mellitus and other categories of glucose intolerance. National Diabetes Data Group. Diabetes. 1979 Dec;28(12):1039-57. doi: 10.2337/diab.28.12.1039. No abstract available. PMID 510803
- [Background] Aburawi EH. The burden of congenital heart disease in libya. Libyan J Med. 2006 Sep 8;1(2):120-2. doi: 10.4176/060902. No abstract available. PMID 21526009